CLINICAL TRIAL: NCT04977297
Title: Move to Music Video Intervention - A Music and Video Guided Exercise Intervention for ICU Survivors
Brief Title: Move to Music Video Intervention for ICU Survivors
Acronym: M2M-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Principal Investigator, Zhan Liang, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201074
Record Dates: First submitted 2021-05-12; First posted 2021-07-26 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Critical Illness; Intensive Care Unit Syndrome
MeSH Terms: conditions — Critical Illness | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move to Music Video Intervention (Experimental): Participants in this arm will receive the Move to Music with Video (M2M-V) intervention. The participant will be asked to exercise twice daily for 5 consecutive days.
  Interventions: Behavioral: Move to Music -Video (M2M-V) Intervention
- Move to Music Intervention (Active Comparator): Participants in this arm will receive the Move to Music (M2M) only intervention without video. The participant will be asked to exercise twice daily for 5 consecutive days.
  Interventions: Behavioral: Move to Music Intervention (M2M)

INTERVENTIONS:
Behavioral: Move to Music Intervention (M2M) — The move to music (M2M) intervention pairs exercise with only music (no video), providing only audio stimulation. The intervention will be provided via an audio playlist that can be played on a phone, tablet, or computer. Each session lasts 10-15 minutes.
  Arms: Move to Music Intervention
Behavioral: Move to Music -Video (M2M-V) Intervention — The move to music video (M2M-V) intervention pairs exercise with both music and video, thus providing both audio and visual stimulation. The intervention will be provided via an audio and video playlist that can be played on a phone, tablet, or computer. Each session lasts 10-15 minutes.
  Arms: Move to Music Video Intervention

SUMMARY:
The purpose of this study is to determine if exercising with a music video program will improve physical functions of patients who have been discharged from an Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old;
2. length of ICU stay >5 days (excludes patients with less comorbidity);
3. recruitment within 48 hours of ICU discharge (standardizes time to begin intervention);
4. able to independently move upper and lower extremities (required to participate in intervention);
5. cognitively able to complete the assessments and comply with physical testing instructions;
6. able to speak English or Spanish; and
7. reside at home prior to ICU admission.

Exclusion Criteria:

1. documented mental incompetence;
2. dependent status pre-ICU admission (assessed by the Katz Index of Independence in Activities of Daily Living);
3. evidence of delirium assessed using the Confusion Assessment Method;
4. hearing impairment;
5. documented "comfort measures only" or impending death;
6. prior residence in a long-term care facility; and
7. unstable clinical measures defined as Heart Rate (>140 beats/minute) or Respiratory Rate (>35 breaths/minute), blood pressure (systolic blood pressure >180 mmHg or < 90mmHg), ventilation problems, agitation, or perspiration. We will not enroll adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in global health | baseline, up to 30 days
  Patient-Report Outcomes Measurement Information System (PROMIS) Global Health is a 10 item questionnaire representing physical health, pain, fatigue, mental health, social health and overall health. The questionnaire has a total score ranging from 10 to 50 with the higher score reflects better functioning.
Change in physical activity | baseline, day5
  Physical activity will be monitored using an Actiwatch (Philips Respironics) placed on subjects' wrists at enrollment. The Actiwatch is a small, lightweight, limb-worn activity monitoring device.
Change in handgrip strength | baseline, up to 30 days
  Handgrip strength will be assessed using handgrip dynamometer.

SECONDARY OUTCOMES:
Number of interventions completed | day 5
  Number of interventions completed will be assessed from self-reported exercise diary.
Patient Satisfaction Survey Scores | day 5
  Participants will complete a Patient Satisfaction survey by rating their experience of using the intervention from 1 to 5 with the higher score indicating a better experience.
Exercise motivation as measured by the Physical Activity Enjoyment Scale | day 5
  The Physical Activity Enjoyment Scale assesses participant's motivation to exercise. The questionnaire has 16 items evaluated on a 7-point Likert Scale. The total score ranges from 16 to 112 with the lower score indicating greater enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhan Liang, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No